CLINICAL TRIAL: NCT06786169
Title: Cohort Studies of Associations of Psychological Stress With Therapy Efficacy and Prognosis of Gastric Cancer (G-STRESS)
Brief Title: The Relationship of Psychological Stress With Therapy Efficacy and Prognosis of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Other Study IDs: G-STRESS
Record Dates: First submitted 2024-09-05; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer
Keywords: Gastric Cancer; Stress
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: advanced gastric cancer patients receiving surgery
  Interventions: Other: psychological stress status
- Cohort 2: stage III-IV gastric cancer patients receiving preoperative treatment
  Interventions: Other: psychological stress status
- Cohort 3: stage IV gastric cancer patients receiving chemotherapy, immunotherapy or ta
  Interventions: Other: psychological stress status

INTERVENTIONS:
Other: psychological stress status — The assessment of depressive and anxiety symptoms was conducted using Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder Assessment 7 (GAD-7). Patients with a PHQ-9 score ≥ 5 or a GAD-7 score ≥ 5 were categorized as the stressed group.

SUMMARY:
This is the prospective, observational cohort study (G-Distress) to explore the associations of psychological stress with treatment and prognosis of gastric cancer. The participants including the patients diagnosed with gastric cancer who received surgery, chemotherapy and immune checkpoint inhibitors.

ELIGIBILITY:
Cohort 1

Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 80 years old, ECOG (ECOG score standard) performance status of 0 or 1
2. Be proven to be primary adenocarcinoma of gastric cancer and staged II-III by pathological evidences
3. R0 gastrectomy with D2 lymphadenectomy
4. Receiving adjuvant chemotherapy

Exclusion Criteria:

1. History of chemotherapy, radiotherapy, immunotherapy or target therapy
2. Multiple primary tumors
3. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases
4. Unavailable for R0 resection and D2 lymph node dissection.
5. Patients with stage IV gastric cancer

Cohort 2

Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 80 years old, ECOG (ECOG score standard) performance status of 0 or 1
2. Be proven to be primary adenocarcinoma of gastric cancer and staged III-IV by pathological evidences
3. Receiving gastrectomy
4. Receiving preoperative chemotherapy

Exclusion Criteria:

1. Unavailable for chemotherapy, radiotherapy, immunotherapy or target therapy
2. Multiple primary tumors
3. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases
4. Unavailable for gastrectomy

Cohort 2

Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 80 years old, ECOG (ECOG score standard) performance status of 0 or 1
2. Be proven to be primary adenocarcinoma of gastric cancer and staged IV by pathological evidences
3. Unavailable for gastrectomy
4. Presence of at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors version 1.1

Exclusion Criteria:

1. Unavailable for chemotherapy, radiotherapy, immunotherapy or target therapy
2. Multiple primary tumors
3. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastric cancer patients
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Disease-free survival (DFS) | 3-year
  The duration between the date after surgery to the date of any recurrence or death firstly
Cohort 2: Pathologic complete response (pCR) rate | 1-month
Cohort 3: Progression-free survival (PFS) | 1-year

SECONDARY OUTCOMES:
Overall survival (OS) | 3-year
Objective Response Rate | through study completion, an average of 1 year
Quality of life assessed by EORTC QLQ-C30. | 3-year

OTHER OUTCOMES:
The correlation between gut microbiota and stress and prognosis | 3-year
The correlation between ctDNA and chronic stress and prognosis | 3-year
The correlation between tumor microenvironment signature and stress and prognosis | 3-year
The correlation between peripheral stress biomarker and immune cells signature and stress and prognosis | 3-year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided